CLINICAL TRIAL: NCT02770027
Title: Impact of Intravascular Fluid Resuscitation on Whole Blood Viscosity During Colon Surgery
Brief Title: Impact of Intravascular Fluid Resuscitation and Whole Blood Viscosity for Colon Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Yop Kim, MD PhD, Professor, Konkuk University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KUH000013
Record Dates: First submitted 2016-05-10; First posted 2016-05-12 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Colon Surgery
Keywords: Colon Surgery; blood viscosity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous Crystalloid (Placebo Comparator): Crystalloid is administered to maintain stroke volume variation < 15 during volume controlled ventilation (8 ml/kg tidal volume) of O2/air mixture
  Interventions: Drug: Intravenous Crystalloid
- Intravenous HES (Active Comparator): HES is administered to maintain stroke volume variation < 15 during volume controlled ventilation (8 ml/kg tidal volume) of O2/air mixture
  Interventions: Drug: Intravenous HES

INTERVENTIONS:
Drug: Intravenous Crystalloid — Crystalloid is administered to maintain stroke volume variation < 15 during volume controlled ventilation (8 ml/kg tidal volume) of O2/air mixture
  Arms: Intravenous Crystalloid
Drug: Intravenous HES — HES is administered to maintain stroke volume variation < 15 during volume controlled ventilation (8 ml/kg tidal volume) of O2/air mixture
  Arms: Intravenous HES

SUMMARY:
After obtaining approval from the Institutional Review Board of our institution, written informed consent is obtained from patients undergoing colon surgery are enrolled in this prospective study and randomly allocated into one of two groups: Group-C (n=15) and Group-HES (n=15).

All recruited patients will be given patient identification number (PIN) for the present study of 01-30 according to their order of interview and recruitment. Investigators will prepare 15 yellow and 15 green cards, which will be inserted in 30 thick-paper envelopes. Then, all envelopes will be sealed, mixed and randomly allocated to get numbers of 01 to 30 (Envelop number).

According to the color of the card, attending anesthesiologists will give crystalloid for yellow card or HES for green cards, respectively, to maintain stroke volume variation < 15 during volume controlled ventilation (8 ml/kg tidal volume) of O2/air mixture.

Patient data and statistical analyses:

Patient's data whole blood viscosity, PaO2, FiO2, Hemoglobin, urine amount, s-glucose will be determined from the patients' medical record after patient's discharge.

All statistical analyses will be performed after the 30th patient's discharge and data acquisition

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing colon surgery
* Patients provided a written informed consent.
* Patients with preoperative serum hemoglobin concentration >13 g/dL (male) and >12 g/dL (female)
* Patients with PaO2/FiO2 ratio >150

Exclusion Criteria:

* Patients with history of anemia, dyspnea, active infection.
* Patients with endocrine disease
* Patients received or receiving intraoperative and preoperative blood salvaged, allogenic blood transfusion, anti-platelet drug, anti-fibrinolytic agents or recombinant human erythropoietin, or undergoing acute normovolemic hemodilution.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
whole blood viscosity | with 1 hour after the completion of procedure
  whole blood viscosity measured by viscometer cm-1

SECONDARY OUTCOMES:
PaO2/FiO2 ratio | 1 hour after the completion of procedure
  PaO2/FiO2 ratio measured by arterial blood gas analysis
hematocrit | 1 hour after the completion of procedure
  serum hematocrit, %
glucose | 1 hour after the completion of procedure
  serum glucose level, g/dl
osmolarity | 1 hour after the completion of procedure
  serum osmolarity, mOsm
urine output | 1 hour after the completion of procedure
  hourly urine output, ml/hr
Maximum clot formation | 1 hour after the completion of procedure
  Maximum clot formation in rotational thromboelastometry (ROTEM) analysis, mm

IPD SHARING:
Plan to Share IPD: No